CLINICAL TRIAL: NCT00427440
Title: A Multicenter, Open-label, Single Agent, Two-stage Phase 2 Study to Evaluate the Efficacy and Safety of AMG 102 in Subjects With Advanced Malignant Glioma
Brief Title: A Phase II Study to Treat Advanced Malignant Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20050253
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Advanced Malignant Glioma
Keywords: Glioma; Brain Tumor
MeSH Terms: conditions — Glioma; Brain Neoplasms

ARMS (2):
- AMG 102 at 10 mg/kg Dose Level (Experimental): Up to 40 subjects will be treated at this dose level based upon investigator assessment of responses observed.
  Interventions: Drug: AMG 102 at 10 mg/kg
- AMG 102 at 20 mg/kg Dose Level (Experimental): Up to 40 subjects will be treated at this dose level based upon investigator assessment of responses observed.
  Interventions: Drug: AMG 102 at 20 mg/kg

INTERVENTIONS:
Drug: AMG 102 at 20 mg/kg — AMG 102 at 20 mg/kg IV (in the vein) every 2 weeks
  Arms: AMG 102 at 20 mg/kg Dose Level
Drug: AMG 102 at 10 mg/kg — AMG 102 at 10 mg/kg IV (in the vein) every 2 weeks
  Arms: AMG 102 at 10 mg/kg Dose Level

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of AMG 102 for the treatment of Advanced Malignant Glioma.

ELIGIBILITY:
Inclusion Criteria:

* subjects with documented histologically confirmed primary grade 4 advanced malignant glioma
* no more than 3 prior relapses or prior systemic treatments
* recurrent disease documented by MRI after prior therapy
* must have at least one site of bidimensionally measurable disease:
* archived tissue from the initial diagnosis of advanced malignant glioma or upon transformation to advanced malignant glioma are available for central review within approximately 4 weeks after enrollment
* age ≥ 18 years
* Karnofsky performance score ≥ 60%
* hemoglobin ≥ 10 g/dL
* absolute neutrophil count ≥ 1.5 x 10(9th)/L
* platelet count ≥ 100 x 10(9th)/L
* serum creatinine ≤ 1.5 times upper limit of normal
* alanine aminotransferase ≤ 2.5 times upper limit of normal
* serum total bilirubin ≤ 2.5 times upper limit of normal
* before any study-specific procedure, the appropriate written informed consent must be obtained

Exclusion Criteria:

* history of central nervous system bleeding as defined by stroke or intraocular bleed (including embolic stroke) within 6 months before enrollment
* evidence of acute intracranial/intratumoral hemorrhage; except for subjects with stable grade 1 hemorrhage
* received radiation therapy within 4 weeks before enrollment or have not recovered from the toxic effects of such therapy
* treated previously with any c-Met or HGF targeted therapy
* treated with thalidomide or tamoxifen within 1 week before enrollment or has not recovered from the toxic effects of such cancer therapy
* treated with immunotherapeutic agents, vaccines or mAb therapy within 4 weeks before enrollment or have not recovered from the toxic effects of such cancer therapy
* treated with alkylating agents within 4 weeks before enrollment or has not recovered from the toxic effects of such cancer therapy
* treated with chemotherapy (non-alkylating agents) within 2 weeks before enrollment or has not recovered from the toxic effects of such cancer therapy
* surgical resection of brain tumor within 4 weeks before enrollment or have not recovered from acute side effects of such therapy, except for neurological effects
* plans to receive surgery, radiation therapy or other elective surgeries during the course of the study
* concurrent severe and/or uncontrolled medical disease (e.g., uncontrolled diabetes, congestive cardiac failure, myocardial infarction within 6 months before enrollment) that could compromise participation in the study
* active infection within 7 days before enrollment
* past or current history of another neoplasm, except for curatively treated non-melanoma skin cancer, carcinoma in situ of the cervix and other primary solid cancer with no known active disease present and no curative or adjuvant treatment administered for the last 3 years
* documented history of human immunodeficiency virus
* documented history of chronic viral hepatitis
* concurrent or prior (within 7 days of enrollment) anticoagulation therapy, except:

  * Use of low molecular weight heparins (LMWH, e.g., enoxaparin sodium [Lovenox] and unfractionated heparin for prophylaxis against central venous catheter thrombosis is allowed
  * Use of low dose warfarin (< 2 mg/day) for prophylaxis against central venous catheter thrombosis is allowed
* currently enrolled in or has not yet completed at least 30 days since ending other investigational device or therapeutic study(s)
* had major surgery within 4 weeks before enrollment or recovering from prior surgery
* known allergy or sensitivity to any of the excipients in the investigational product
* pregnant or breast feeding
* unwilling to use adequate contraceptive precautions during the course of the study and for 6 months after the last administration of investigational product, for:

  * male subjects
  * female subjects who are not post-menopausal (no menstrual period for a minimum of 12 months at study entry) or documented surgically sterile will not be bound to this exclusion
* previously treated with AMG 102
* previously enrolled into this study
* will not be available for follow-up assessment
* has other disorders that compromises the ability of the subject to give written informed consent and/or comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2006-11; Primary Completion 2008-12 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Assess best objective confirmed response rate in subjects with advanced malignant glioma receiving AMG 102 treatment | Week 9 from first dose of AMG 102

SECONDARY OUTCOMES:
To assess the safety profile of AMG 102 in subjects with advanced malignant glioma | entire study
Estimate overall survival and progression-free survival rates in this population | 8 week intervals
Assess the duration of response and time to response in this population | Treatment Period
Assess the pharmacokinetics of AMG 102 in subjects with advanced malignant glioma | Weeks 1, 5, and 9

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Wen PY, Schiff D, Cloughesy TF, Raizer JJ, Laterra J, Smitt M, Wolf M, Oliner KS, Anderson A, Zhu M, Loh E, Reardon DA. A phase II study evaluating the efficacy and safety of AMG 102 (rilotumumab) in patients with recurrent glioblastoma. Neuro Oncol. 2011 Apr;13(4):437-46. doi: 10.1093/neuonc/noq198. Epub 2011 Feb 4. PMID 21297127
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com